CLINICAL TRIAL: NCT02002689
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module - 5 LDE225 for Patients With PTCH1 or SMO Mutated Tumors
Brief Title: LDE225 for Patients With PTCH1 or SMO Mutated Tumors
Acronym: SIGNATURE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225XUS20
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: PTCH1 or SMO Activated Solid and Hematologic Tumors
Keywords: Solid tumor malignancy,; hematologic malignancy,; mutation, translocations,; signature,; PTCH1,; SMO,; LDE225,; endometrial cancer,; colon cancer,; bladder,; NSCLC
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Hematologic Neoplasms; Endometrial Neoplasms; Colonic Neoplasms | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDE225 (Experimental): LDE225 800 mg (hard gelatin capsules) will be administered orally once daily on a continuous dosing schedule.
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — LDE225 800 mg (hard gelatin capsules) will be administered orally once daily on a continuous dosing schedule

SUMMARY:
The purpose of this signal seeking study is to determine whether treatment with LDE225 demonstrates sufficient efficacy in hedgehog pathway-mutated solid tumors and/or hematologic malignancies to warrant further study

ELIGIBILITY:
Inclusion Criteria:

* Patient has confirmed diagnosis of a select solid tumor (except medulloblastoma, basal cell carcinoma and pancreatic adenocarcinoma) or hematological malignancy (except CML, ALL and AML).
* Patient has pre-identified tumor with a PTCH1 or SMO mutation.
* Patient has received at least one prior treatment for recurrent, metastatic and /or locally advanced disease and for whom no standard therapy options are anticipated to result in a durable remission.
* Patient has progressive and measurable disease as per RECIST 1.1. or other appropriate hematological guidelines.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

* Patients has received prior treatment with LDE225.
* Patients has neuromuscular disorders associated with elevated CK (i.e. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis
* Patients has primary CNS tumor or CNS tumor involvement
* Patient has received chemotherapy or anticancer therapy ≤ 4 weeks prior to starting study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California Davis Cancer Center UC Davis Cancer (3), Sacramento, California
  - Rocky Mountain Cancer Centers RMCC - Aurora, Greenwood Village, Colorado
  - Lurie Children's Hospital of Chicago Developmental Therapeutics, Chicago, Illinois
  - Minnesota Oncology Hematology, P.A. Southdate Medical Center, Minneapolis, Minnesota
  - Cleveland Clinic Foundation Cleveland Clinic (19), Cleveland, Ohio
  - Sanford Research Sanford Health, Sioux Falls, South Dakota
  - Oncology Consultants Oncology Group, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (3), Houston, Texas
  - Intermountain Medical Center Intermountain Healthcare, Murray, Utah
  - Seattle Cancer Care Alliance Skagit Valley Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was closed for accrual when the sponsor realized that not enough patients will be recruited for any meaningful stat analysis even if the study were kept open beyond the original planned accrual window.
Groups:
- Sonidegib: All the patients received sonidegib on a flat scale of 800 mg (e.g., 4 x 200 mg hard gelatin capsules) once daily on a continuous dosing cycle.
Period: Overall Study
Arm/Group | Sonidegib
Started | 10
Completed | 0
Not Completed | 10
Not completed — Disease Progression | 7
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sonidegib
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Summary of Overall Response (ORR) and Clinical Benefit (CBR)
Description: Clinical benefit rate (CBR) Number and percentage of subjects with CBR (responses of CR, PR or SD ≥ 16 weeks) as assessed by investigator was reported for all patients along with 95% exact confidence interval (CI). Overall Response Rate (ORR) Overall response was to be determined by investigator assessment for each tumor in the study. For subjects with solid tumors, the assessment criteria was RECIST 1.1 and included responses of CR and/or PR. The number and percentage of subjects for different categories of overall response (e.g., for solid tumors - CR, PR, SD, PD, Not Evaluable) were to be provided for solid tumors, and each hematological tumor type (if applicable). Ninety-five percent (95%) exact CI was to be provided for the response rate(s) (e.g., for solid tumors - CRn and/or PR) as well.
Time Frame: 16 weeks
Population: Full analysis set
Measure: Number; unit: percent responders
Arm/Group | Sonidegib
Number analyzed (Participants) | 10
percent responders
  Complete response (CR) | 0
  Partial response (PR) | 0
  Stable disease (SD) | 0
  Progressive disease (PD) | 8
  Non-evaluable (NE) | 2
  Overall response rate (ORR: CR+PR) | 0
  Clinical benefit rate (CBR: CR+PR+SD) | 0

2. Secondary Outcome: Summary of Timing and Estimated Rate for Progression-free Survival (PFS) - Full Analysis Set
Description: Progression-free survival (PFS) is the time from the date of start of treatment to the date of event defined as the first documented progression or death due to any cause within 30 days of last dose. If a subject has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
Time Frame: 4 months
Population: Full Analysis set
Measure: Number (95% Confidence Interval); unit: % progression free surviors
Arm/Group | Sonidegib
Number analyzed (Participants) | 10
% progression free surviors
  1 Month | 88.9 [43.3 to 98.4]
  2 Months | 33.3 [7.8 to 62.3]
  3 Months | 33.3 [7.8 to 62.3]
  4 Months | 0.0 [NA to NA] — limits not needed for 0 observations

3. Secondary Outcome: Kaplan-Meier Estimates of Progression Free Survival (PFS )Timing, Months
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sonidegib
Number analyzed (Participants) | 10
months | 1.8 [0.9 to 3.6]

ADVERSE EVENTS:
Groups:
- LDE225: All the patients received sonidegib on a flat scale of 800 mg (e.g., 4 x 200 mg hard gelatin capsules) once daily on a continuous dosing cycle.
Arm/Group | LDE225
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 (N=10)
Abdominal pain (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 (N=10)
Anaemia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Fatigue (General disorders) | 6
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 3
Haemoglobin decreased (Investigations) | 1
Weight decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
The study was closed for accrual when the sponsor realized that not enough patients will be recruited for any meaningful stat analysis even if the study were kept open beyond the original planned accrual window.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary.

However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.